CLINICAL TRIAL: NCT06399081
Title: A Real-world Study of Predictive Models of Gangrenous Cholecystitis Based on Machine Learning
Brief Title: Construction of a Predictive Model of Gangrenous Cholecystitis Based on Machine Learning
Status: Completed | Type: Observational
Sponsor: Dalian Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Ying Ma, resident physician, Dalian Medical University
Other Study IDs: KY2024-006-02
Record Dates: First submitted 2024-04-29; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Gangrenous Cholecystitis
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gangrenous cholecystitis: Defined based on intraoperative findings or pathological diagnosis
  Interventions: Other: Observational
- Non-gangrenous cholecystitis: Non-gangrenous cholecystitis, such as chronic cholecystitis, acute cholecystitis, acute attack of chronic cholecystitis
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
Gangrenous cholecystitis is the most common complication of acute cholecystitis.

There is no research using machine learning models to construct predictive diagnostic models for gangrenous cholecystitis.

DETAILED DESCRIPTION:
This study reviewed the clinical data of 2023 cholecystectomy patients admitted to our center between January 1, 2015, and May 31, 2015, it includes demographic, clinical features, laboratory and imaging indexes, and constructs five commonly used Decision Tree, SVM, Random Forest, XGBoost, AdaBoost models, feature subsets are selected by Recursive Feature Elimination with Cross-Validation and the importance of variables in each model, model performance is evaluated by Balanced accuracy, Recall, Precision, F1score, and the Precision-Recall(PR) curve, and the final results are verified by independent external validation sets.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with acute cholecystitis or acute exacerbation of chronic cholecystitis in our hospital and receiving complete clinical treatment in our hospital;
* performing cholecystectomy;
* having complete and searchable clinical data, such as patient's age, surgical records, and hospitalization days.

Exclusion Criteria:

* previous diagnosis of chronic cholecystitis, this time for elective surgical treatment;
* previous diagnosis of acute cholecystitis, ultrasound-guided cholecystectomy after elective laparoscopic cholecystectomy;
* concomitant with other acute biliary and pancreatic system-related diseases, such as obstructive jaundice caused by choledochal stones, acute cholangitis, acute pancreatitis, etc.;
* exclude patients who combined with other surgery patients such as choledochotomy and lithotripsy, choledochoscopic exploration and lithotripsy, bile-intestinal anastomosis, appendectomy, etc;
* those with incomplete data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients admitted to the Second Hospital of Dalian Medical University who were diagnosed with cholecystitis through ICD-9 code recognition and underwent cholecystectomy from January 2015 to May 2023
Sampling Method: Non-Probability Sample
Enrollment: 1006 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
pathological diagnosis of patients with cholecystectomy | 30 days
  Check the patient's pathological report and whether the pathological description contains phenomena such as full layer ischemic necrosis and ulceration of the gallbladder wall. Diagnose as gangrenous cholecystitis or non-gangrenous cholecystitis.
The predictive performance of diagnostic prediction models | through study completion, an average of 4 months
  The predictive diagnosis was obtained by the model and each predictive variable, and the metric (Accuracy, Recall, Precision, F1score) of the model was obtained by comparing with the actual pathological diagnosis.

SECONDARY OUTCOMES:
WBC value (10*9/L) | through study completion, an average of 4 months
  Correlation between WBC and patients with gangrenous cholecystitis and non-gangrenous cholecystitis
Alanine transaminase value (ALT, U/L) | through study completion, an average of 4 months
  Correlation between liver function and patients with gangrenous cholecystitis and non-gangrenous cholecystitis
D-dimer value | through study completion, an average of 4 months
  Correlation between coagulopathy and patients with gangrenous cholecystitis and non-gangrenous cholecystitis
Fibrinogen value (g/L) | through study completion, an average of 4 months
  Correlation between coagulopathy and patients with gangrenous cholecystitis and non-gangrenous cholecystitis
BMI (Kg/m2) | through study completion, an average of 4 months
  Correlation between obesity level and patients with gangrenous cholecystitis and non-gangrenous cholecystitis
Gallbladder wallness (cm) | through study completion, an average of 4 months
  Correlation between Gallbladder wallness and patients with gangrenous cholecystitis and non-gangrenous cholecystitis

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No
The data where our results derived from were from the Second Hospital of Dalian Medical University. The original data were not publicly available and could only be shared with the permission of the Ethics Committee of the Second Hospital of Dalian Medical University.

REFERENCES:
- [Background] Wu B, Buddensick TJ, Ferdosi H, Narducci DM, Sautter A, Setiawan L, Shaukat H, Siddique M, Sulkowski GN, Kamangar F, Kowdley GC, Cunningham SC. Predicting gangrenous cholecystitis. HPB (Oxford). 2014 Sep;16(9):801-6. doi: 10.1111/hpb.12226. Epub 2014 Mar 17. PMID 24635779
- [Background] Yacoub WN, Petrosyan M, Sehgal I, Ma Y, Chandrasoma P, Mason RJ. Prediction of patients with acute cholecystitis requiring emergent cholecystectomy: a simple score. Gastroenterol Res Pract. 2010;2010:901739. doi: 10.1155/2010/901739. Epub 2010 Jun 8. PMID 20631896
- [Background] Borzellino G, Sauerland S, Minicozzi AM, Verlato G, Di Pietrantonj C, de Manzoni G, Cordiano C. Laparoscopic cholecystectomy for severe acute cholecystitis. A meta-analysis of results. Surg Endosc. 2008 Jan;22(1):8-15. doi: 10.1007/s00464-007-9511-6. Epub 2007 Aug 18. PMID 17704863